CLINICAL TRIAL: NCT02113280
Title: Randomised Controlled Trial Comparing Arthroscopy With Physiotherapy for Degenerative Meniscal Tears
Brief Title: DEMAND - DEgenerative Meniscal Tears - Arthroscopy vs. Dedicated Exercise
Acronym: DEMAND
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed funding application.
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Sarah Johnson-Lynn, Specialty Registrar, Northumbria Healthcare NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUTH-DJK-2013
Record Dates: First submitted 2013-10-16; First posted 2014-04-14 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Degenerative Meniscal Tears; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroscopy; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapy (Active Comparator): Physiotherapy
  Interventions: Procedure: Physiotherapy
- Arthroscopy (Experimental): Arthroscopy
  Interventions: Procedure: Arthroscopy

INTERVENTIONS:
Procedure: Arthroscopy — Patients to receive knee arthroscopy and meniscal debridement
  Arms: Arthroscopy
Procedure: Physiotherapy — Outpatient standardised physiotherapy regime with focus on exercise therapy
  Arms: Physiotherapy

SUMMARY:
Patients with wear and tear in their knees (osteoarthritis) are often referred to orthopaedic surgeons following a sudden worsening of pain and mechanical symptoms (grinding, locking, giving way) in their knee due to tears of their meniscal cartilages. These tears are described as degenerative as they are not usually caused by a single injury but rather accumulation of wear and tear. It is not clear from the current available evidence what the best treatment for these patients is. Their underlying arthritis is not bad enough to require joint replacement yet and they were usually managing well with minimal problems from their knee until experiencing the meniscal tear. However, some of their symptoms are likely to be due to the arthritis rather than just the tear. Current treatment for these patients is usually in the form of conservative treatment with physiotherapy and supervised exercise or using arthroscopy (key-hole surgery) to trim the damaged area of the meniscus. We know from previous research that most of these patients will improve over time to some extent but it is not clear whether a greater improvement can be expected following surgery and if so, whether this applies to all patients with this problem or not.

Our study is intended to compare the outcome of patients with proven degenerative meniscal tears imaged on MRI scans, when they are assigned to arthroscopy followed by supervised exercise or supervised exercise alone. They will be randomly assigned and the outcome will be assessed using patient-completed questionnaires (Knee Outcome Osteoarthritis and injury Score [KOOS], SF12, visual analogue score for pain) and whether the patients go on to require further surgery during the period of the trial. The patients will be assessed at baseline, at 6 weeks, 6 months, 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age over 45 years
* Knee pain in the presence of a medial meniscal tear on MRI.

Exclusion Criteria:

* History of trauma to the knee or ipsilateral lower limb in the past 2 years
* Inability to engage in postoperative rehabilitation
* Lacking capacity to consent
* Evidence of infection
* Previous knee surgery other than arthroscopy (diagnostic or partial meniscectomy) Neurological disease
* Inflammatory arthritis
* Loose bodies
* Ligament injuries causing symptomatic instability
* Women who are pregnant
* Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* Uncontrolled disease states, such as moderate/severe asthma, COPD or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids, or recurrent infections.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Knee injury and Osteoarthritis Outcome Score | 6weeks, 6 months, 12 months, 24 months
  Patient completed outcome measure

SECONDARY OUTCOMES:
SF12 | 6 weeks, 6 months, 12 months, 24 months
  Patient completed outcome measure
Pain visual analogue score | 6 weeks, 6 months, 12 months, 24 months
  Patient completed outcome measure

CONTACTS AND LOCATIONS:
Locations (1):
- North Tyneside General Hospital, North Shields, Tyne and Wear, United Kingdom